CLINICAL TRIAL: NCT02878174
Title: The Site of Puncture in Ultrasound-guided Prelocation Technique of the Internal Jugular Venous Catheterization: Non-inferiority Randomized Clinical Trial
Brief Title: The Site of Puncture in Prelocation Technique of the Internal Jugular Venous Catheterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IJV_rotation
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Jugular Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional ultrasound (US)-guided group (Active Comparator): internal jugular vein catheterization using conventional US-guided internal jugular vein (IJV) cannulation
  Interventions: Procedure: internal jugular vein catheterization
- rotational Prelocation group (Experimental): internal jugular vein catheterization using landmark approach based on the rotation-adjusted US screen
  Interventions: Procedure: internal jugular vein catheterization

INTERVENTIONS:
Procedure: internal jugular vein catheterization — internal jugular vein catheterization using ultrasound (US) or US-based prelocation techniques

SUMMARY:
Two approaches such as ultrasound (US)-guided and prelocation techniques are possible when the internal jugular vein cannulation is attempted with US. This study is a clinical trial that compares the success rates of both techniques and shows the non-inferiority of the prelocation technique. However, during prelocation technique, rotated screen of the US is used instead of original screen. The angle of rotation is determined by the degree of rotation of US probe where an accelerometer is attached.

DETAILED DESCRIPTION:
The investigator's own developed screen-rotating program is used. An accelerometer is attached on the front surface of the ultrasound (US) probe. The angle of rotation of the probe is delivered to the laptop and becomes the information to adjust the rotating angle of screen. Immediately after induction of general anesthesia, the patient's head is turned slightly, and the table is tilted at 10 degrees. In the US group, the investigators obtain a sonographic view and try a cannulation of the internal jugular vein (IJV). In the prelocation group, a skin marker is made on the anticipated skin puncture site where a perpendicular line that passes over the center of the IJV meets the skin on the rotated US screen. It is recorded "success" when the internal jugular vein is successfully punctured without complications. It is recorded "failure" if the internal jugular vein is not punctured during repeated needle passes. The number of tries and tile to success are recorded. The success and complication rates between two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anesthesia

Exclusion Criteria:

* Refusal of consent
* Patients with cervical spine injuries
* Patients with atlanto-axial instability
* Patients at risk of increased intracranial pressure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of internal jugular vein cannulation | intraoperative

SECONDARY OUTCOMES:
Degree of rotation of ultrasound (US) probe | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No